CLINICAL TRIAL: NCT03377920
Title: Predictive Value of Peak Inspiratory Flow Rate Derived From Spirometry to Determine the Patient's Ability to Produce Peak Inspiratory Flow Rate to Overcome the Resistance of Current Dry Powders Inhalers.
Brief Title: Predictive Value of Spirometric PIF to Produce PIF Rate Needed for the Use of Current DPI's.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 143201733083
Record Dates: First submitted 2017-10-26; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-10

CONDITIONS: Severe Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe asthma patients; COPD patients (Experimental): Cross sectional study Lung function measurement
  Interventions: Device: In-check Dial device (Clement Clarke International Ltd, Harlow, UK)

INTERVENTIONS:
Device: In-check Dial device (Clement Clarke International Ltd, Harlow, UK) — * pre-bronchodilator spirometry for the measurement of PIFspiro as per ERS/ATS guidelines for standard lung function5 (part of routine clinical follow-up).
  * 5 forced inspiratory manoeuvres using the In-check Dial device G16, set at 5 different resistances (performed in order of increasing resistance), yielding the PIFresist values for the different DPI's

SUMMARY:
The main aim is to study correlations between Peak inspiratory flow measured during a spirometry (PIFspiro) and Peak inspiratory flow measured over a pre-set resistance (PIFresist) in COPD patients and severe asthma patients. PIFresist will be measured using 5 different resistances, representing all DPI's relevant for the treatment of obstructive lung diseases. If this shows a distinct relationship between PIFspiro and PIFresist, PIFspiro cut-off points will be sought in an attempt to predict which patients are likely to be able to produce optimal flows for DPI use. If successful, this will make the actual measurement of PIFresist redundant in clinical practice. Also the relationship between PIFresist and device internal resistance in addition to PIFspiro (which corresponds to a very low resistance) will be examined.

DETAILED DESCRIPTION:
The correct use of dry powder inhalers (DPI) crucially depends on the peak inspiratory flow (PIF) that the patient can generate when overcoming internal resistance of the inhaler device.

It has been shown that some patients cannot achieve sufficient peak inspiratory flows with some DPI's, especially in the elderly population. The In-check Dial device (Clement Clarke International Ltd, Harlow, UK) allows to measure these inspiratory flows for different pre-set resistances, representing different DPI's.

Study design: interventional, single center, single visit study

30 Severe asthmatics and 70 COPD patients will be recruited in the UZ Brussel respiratory outpatient clinic.

All participants will provide written informed consent.

Patients will perform:

* pre-bronchodilator spirometry for the measurement of PIFspiro as per European respiratory Society/American Thoracic Society (ERS/ATS) guidelines for standard lung function5 (part of routine clinical follow-up).
* 5 forced inspiratory manoeuvres using the In-check Dial device G16, set at 5 different resistances (performed in order of increasing resistance), yielding the PIFresist values for the different DPI's

ELIGIBILITY:
Inclusion Criteria:

* Severe asthmatics (M/F; > 20 y) entering the Belgian Severe Asthma Registry (BSAR)
* COPD patients (GOLD stage II-IV; M/F; > 40 y)

Exclusion Criteria:

* Inability to perform spirometry

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
PIFspiro | At inclusion (D0)
  PIFspiro (L/s): PIF measurement from standardized spirometry (3 flow-volume measurements);
PIFresist | At inclusion (D0)
  PIFresist (L/min): PIF from In-check Dial (5 flow measurements with flow restrictor in 5 different positions)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Hanon, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No